CLINICAL TRIAL: NCT01346241
Title: Improving Access To Services With An Intensive Two-Day Treatment For Panic
Brief Title: Improving Access To Services to Community Based Outpatient Clinics (CBOC's)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Ellen Teng, Ph.D, Michael E. DeBakey VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-28272
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Panic Disorder
Keywords: Panic; Anxiety
MeSH Terms: conditions — Panic Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Intensive Panic Control Treatment (IPCT) — A manualized treatment that consists of psychoeducation about panic disorder
  Other Names: Panic Disorder

SUMMARY:
The purpose of this study is to examine the feasibility of delivering IPCT in three rural VA community based outpatient clinics (CBOCs).

DETAILED DESCRIPTION:
We will first need to develop a more thorough understanding of the potential barriers associated with implementing this novel form of treatment in these settings by conducting focus groups at each facility. This information will then be used to modify the treatment, which will then be piloted with Veterans enrolled in these clinics who have panic disorder.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF/OND Veteran with current diagnosis of panic disorder with or without agoraphobia (presence of other anxiety disorders is acceptable)

Exclusion Criteria:

* Current substance dependence
* psychosis
* symptomatic bipolar disorder
* severe depression with suicidal intent or plan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Intensive Panic Control Treatment (IPCT) | 3 Months
  IPCT is a manualized treatment that consists of psychoeducation about panic disorder, behavioral exercises such as breathing retraining and interoceptive exposure to mimic symptoms during an actual panic attack, and cognitive restructuring (identifying thought distortions and replacing them with corrective thoughts based on realistic appraisals).

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Teng, Ph.D, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. DeBakey VA Medical Center and CBOC's (Lufkin, Texas City, and Conroe), Houston, Texas, United States